CLINICAL TRIAL: NCT01063140
Title: Rabies Immune Plasma Booster Program - A Clinical Study Conducted as an Investigational New Drug Study
Brief Title: Rabies Immune Plasma Booster Study
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Collaborators: CSL Plasma (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZLB 1
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Rabies
Keywords: Rabies Immune Globulin; Source Plasma Donors; Booster Immunization
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- RabAvert
  Interventions: Biological: Rabies Vaccine (RabAvert)
- Imovax
  Interventions: Biological: Rabies Vaccine (Imovax)

INTERVENTIONS:
Biological: Rabies Vaccine (RabAvert) — The initial booster immunization is given on Day 1; subsequent booster immunizations will be administered if the donor's titers fall below 10 IU/mL. A maximum of 4 booster immunizations may be administered over the 2 year study period.
  Other Names: Rabipur
  Groups: RabAvert
Biological: Rabies Vaccine (Imovax) — The initial booster immunization is given on Day 1; subsequent booster immunizations will be administered if the donor's titers fall below 10 IU/mL. A maximum of 4 booster immunizations may be administered over the 2 year study period.
  Groups: Imovax

SUMMARY:
Rabies immune globulin is a product that is lifesaving to unvaccinated individuals exposed to the rabies virus. Rabies immune globulin is made from plasma from immune donors. Currently the only practical method to obtain this plasma is to immunize normal volunteer Source Plasma donors and collect their plasma while titers are adequate. The use of rabies vaccine for immunization of normal Source Plasma donors is currently limited to a level that, while protective for the individual, is unsuitable for production of rabies immune globulin.

The objective of this study is to obtain efficacy and safety data regarding the rabies boostering program to demonstrate that:

1. Rabies immune plasma production can be substantially increased by giving booster doses to previously immunized donors whose titers are below 10.0 IU/mL.
2. It is safe for normal Source Plasma donors to receive booster doses of rabies vaccine on a regular basis.

This study utilizes two rabies vaccines approved by the FDA, Imovax® (Sanofi-Pasteur) and RabAvert® (Novartis).

ELIGIBILITY:
Inclusion Criteria:

* Meet requirements for Source Plasma donors
* Completed initial series of rabies antibody injections with no serious adverse events for at least 90 days prior to enrollment
* Compliance with program requirements
* Signed informed consent

Exclusion Criteria:

* Failure to meet requirements to be Source Plasma donor
* Non-compliance with the program
* Experience a serious adverse reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Source Plasma Donors. Donors must meet FDA and CSL Plasma requirements to be Source Plasma Donors. Donors had previously participated in CSL's rabies vaccine immunization program.
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) for rabies plasma donations received after booster injections | 30-day intervals for the duration of the study (up to 2 years)

SECONDARY OUTCOMES:
Adverse Event Reaction Rate | 30-35 days after each injection

CONTACTS AND LOCATIONS:
Overall Officials: Toby L. Simon, MD, Principal Investigator — CSL Plasma
Locations (10):
- United States (10):
  - CSL Donor Plasma Center, Tempe, Arizona
  - CSL Donor Plasma Center, Rock Island, Illinois
  - CSL Donor Plasma Center, Oak Park, Michigan
  - CSL Donor Plasma Center, Saint Paul, Minnesota
  - CSL Donor Plasma Center, Cleveland, Ohio
  - CSL Donor Plasma Center, Springfield, Ohio
  - CSL Donor Plasma Center, Oklahoma City, Oklahoma
  - CSL Donor Plasma Center, Medord, Oregon
  - CSL Donor Plasma Center, Knoxville, Tennessee
  - CSL Donor Plasma Center, Salt Lake City, Utah